CLINICAL TRIAL: NCT02265744
Title: A Phase 2, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Lulizumab Pegol vs. Placebo on a Background of Limited Standard of Care in the Treatment of Subjects With Active Systemic Lupus Erythematosus
Brief Title: Safety and Efficacy Study of a Biologic to Treat Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IM128-027; 2014-002184-14 (EudraCT Number)
Record Dates: First submitted 2014-10-15; First posted 2014-10-16 (Estimated); Results first posted 2019-01-04 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Lupus
MeSH Terms: interventions — lulizumab pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Experimental:Arm A: BMS-931699 (Experimental): 12.5mg subcutaneous (SC) injection Weekly dosing
  Interventions: Drug: BMS-931699
- Experimental:Arm B: BMS-931699 (Experimental): 12.5mg SC injection Every other Week dosing
  Interventions: Drug: BMS-931699
- Experimental:Arm C: BMS-931699 (Experimental): 5mg SC injection Every other Week dosing
  Interventions: Drug: BMS-931699
- Experimental:Arm D: BMS-931699 (Experimental): 1.25mg SC injection Every other Week dosing
  Interventions: Drug: BMS-931699
- Placebo Comparator: Arm E: Placebo matching BMS-931699 (Placebo Comparator): 0mg SC injection Weekly dosing
  Interventions: Drug: Placebo matching BMS-931699

INTERVENTIONS:
Drug: BMS-931699
  Other Names: lulizumab pegol
  Arms: Experimental:Arm A: BMS-931699; Experimental:Arm B: BMS-931699; Experimental:Arm C: BMS-931699; Experimental:Arm D: BMS-931699
Drug: Placebo matching BMS-931699
  Arms: Placebo Comparator: Arm E: Placebo matching BMS-931699

SUMMARY:
Study evaluating the safety and efficacy of a novel biologic in the treatment of systemic lupus erythematosus in male and female adults. Patients who qualify will be randomized to either active BMS-931699 or placebo for initially, up to 24 weeks. Patients who complete the initial 24 weeks of treatment and who are responding to therapy will have the option to continue receiving BMS-931699 as part of a long-term extension (LTE). Disease activity and safety will be assessed over the course of the study through laboratory values, various rating scales accepted in systemic lupus erythematosus studies and patient self reporting.

DETAILED DESCRIPTION:
1. Subjects completing Day 169 (24 weeks) on study medication may be eligible to enter an optional LTE period
2. The LTE period will remain blinded but will no longer have a placebo arm:

   * Subjects will remain on their originally assigned treatment arm unless they were on placebo
   * Subjects initially randomized to placebo arm will be automatically re-randomized into one of the existing active arms at Day 169 (24 weeks)

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Male or female aged between 18 to 70 (included)
* Diagnosed with active systemic lupus erythematosus by a doctor
* Disease must be in patient's joints or on the skin at a minimum
* Taking other medications is allowed but some are excluded

Exclusion Criteria:

* Diagnosed with active lupus nephritis, multiple sclerosis or rheumatoid arthritis
* Diagnosed with active tuberculosis or an ongoing infection with a bacteria or a virus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2014-11-13 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (119):
- United States (25):
  - Rheumatology Associates Of North Alabama, P.C., Huntsville, Alabama
  - St Jude Hospital Yorba Linda, Fullerton, California
  - Valerius Med Group & Res Ctr Of Greater Long Beach, Inc., Long Beach, California
  - Harbor UCLA Medical Center, Torrance, California
  - University Of Connecticut Health Center, Farmington, Connecticut
  - Local Institution, Trumbull, Connecticut
  - Center For Rheumatology, Immunology And Arthritis, Fort Lauderdale, Florida
  - The Arthritis Center, Palm Harbor, Florida
  - Jefrey D. Lieberman, Md., Pc, Decatur, Georgia
  - Coeur D'Alene Arthrit Clin, Coeur d'Alene, Idaho
  - Heartland Research Associates, Llc, Wichita, Kansas
  - Beth Israel Deaconess Med. Center Div. Of Gastroenterology, Boston, Massachusetts
  - Physician Research Collaboration, Llc, Lincoln, Nebraska
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - North Shore Lij Health System, Great Neck, New York
  - The Feinstein Institute For Medical Research, Manhasset, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Joint and Muscle Medical Care and Research Institute (JMMCRI), Charlotte, North Carolina
  - Pmg Research Of Salisbury, Salisbury, North Carolina
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - East Penn Rheumatology Associates, P.C., Bethlehem, Pennsylvania
  - Allegheny-Singer Research Institute (Asri), Pittsburgh, Pennsylvania
  - Tekton Research Inc, Austin, Texas
  - Local Institution, Dallas, Texas
  - Arthritis Northwest, Spokane, Washington
- Argentina (6):
  - Local Institution, Capital Federal, Buenos Aires
  - Hospital General De Agudos J.M. Ramos Mejia, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Instituto De Investigaciones Clinicas De Mar Del Plata, Mar del Plata, Buenos Aires
  - Instituto de Asistencia Reumatologica Integral, San Fernando, Buenos Aires
  - Clinica De Reumatologia, Rosario, Santa Fe Province
  - Centro Consultora Integral de Salud SRL, Córdoba
- Brazil (8):
  - Servicos Especializados em Reumatologia SER, Savaldor, Estado de Bahia
  - Cip Pesquisas Medicas, Goiânia, Goiás
  - Centro Mineiro De Pesquisa, Juiz de Fora, Minas Gerais
  - Centro Medico Varginha, Varginha, Minas Gerais
  - Edumed - Educacao em Saude S/S LTDA, Curitiba, Paraná
  - LMK Servicos Medicos S S Ltda, Porto Alegre, Rio Grande do Sul
  - CPCLIN Centro de Pesquisas Clinicas LTDA, São Paulo
  - Lar Escola AACD, São Paulo
- Canada (5):
  - Karma Clinical Trials Inc., St. John's, Newfoundland and Labrador
  - McMaster University, Hamilton, Ontario
  - Toronto Western Hospital, University Health Network, Toronto, Ontario
  - CHU de Quebec Research Centre, Québec, Quebec
  - Centre De Recherche Musculo-Squelettique, Trois-Rivières, Quebec
- Chile (2):
  - Centro De Estudios Reumatologicos, Santiago, Santiago Metropolitan
  - Hospital San Borja Arriaran, Santiago, Santiago Metropolitan
- Colombia (4):
  - Riesgo De Fractura, Bogota, Cundinamarca
  - Servimed E.U, Bucaramanga, Santander Department
  - Clinica De La Costa, Barranquilla
  - Hospital Pablo Tobon Uribe, Medellín
- France (5):
  - Local Institution, Bordeaux
  - Local Institution, Lille
  - Local Institution, Marseille
  - Local Institution, Paris
  - Local Institution, Strasbourg
- Germany (4):
  - Campus Charite Mitte, Berlin
  - Medizinsche Universitaetsklinik Freiburg, Freiburg im Breisgau
  - Universitaetshautklinik Heidelberg, Heidelberg
  - Johannes Gutenberg - Universitaet, Mainz
- Hungary (3):
  - Budai Irgalmasrendi Korhaz, Budapest
  - Infektologiai-Hepatologiai Osztaly, Gyula
  - Borgyogyaszati Klinika, Szeged
- Italy (5):
  - Arcispedale S. Anna, Cona - Ferrara
  - Azienda Ospedaliera Luigi Sacco, Milan
  - Azienda Ospedaliera Di Padova, Padua
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Policlinico Umberto I, Roma
- Japan (14):
  - Local Institution, Chiba, Chiba
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Kitakyushu-shi, Fukuoka
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Kanazawa, Ishikawa-ken
  - Local Institution, Sendai, Miyagi
  - Local Institution, Sasebo-shi, Nagasaki
  - Local Institution, Shimotsuke-shi, Tochigi
  - Local Institution, Bunkyo-ku, Tokyo
  - Local Institution, Chuo-ku, Tokyo
  - Local Institution, Fuchū, Tokyo
  - Local Institution, Itabashi-ku, Tokyo
  - Local Institution, Meguro-ku, Tokyo
  - Local Institution, Shinjuku-Ku, Tokyo
- Lebanon (2):
  - Local Institution, Beirut
  - Local Institution, Tripoli
- Mexico (9):
  - CINTRE - Centro de investigacion y tratamiento reumatologico, S.C., Mexico City, Distrito Fededral
  - Consultorio Medico de Reumatologia Dr.Jesus Alberto Lopez Garcia, León, Guanajuato
  - Clinica de Investigacion en Reumatologia y Obesidad S.C., Guadalajara, Jalisco
  - Centro Integral En Reumatologia Sa De Cv, Guadalajara, Jalisco, Jalisco
  - Instituto para el DeSarrollo Integral de la Salud S de RL de CV, Mexico City, Mexico City
  - Centro de Radiodiagnostico Computarizado Medico de Tabasco S.A. de C.V., Villahermosa, Tabasco
  - Instituto Nacional De Ciencias Medicas Y Nutricion S.Z., Distrito Federal
  - Centro de Alta Especialidad en Reumatologia e Investigacion del Potosi S.C., San Luis Potosí City
  - Unidad Reumatologica Las Americas, S.C. P., Yucatán
- Netherlands (2):
  - Local Institution, Groningen
  - Local Institution, The Hague
- Peru (3):
  - Clinica Anglo Americana, Lima
  - Hospital Nacional Cayetano Heredia, Lima
  - Instituto De Ginecologia Y Reproduccion Inv. Clinical Sac, Lima
- Poland (3):
  - Local Institution, Lublin
  - Medyczne Centrum Hetmanska Indywidualna Spec. Praktyka Lekar, Poznan
  - Local Institution, Warsaw
- Local Institution, San Juan, Puerto Rico
- Romania (2):
  - Sf. Maria Clinical Hospital,Bucharest, Bucharest
  - Spitalul Clinic de Recuperare Iasi, Iași
- Russia (2):
  - Local Institution, Saint Petersburg
  - Local Institution, Tolyatti
- South Africa (4):
  - Local Institution, Johannesburg, Gauteng
  - Local Institution, Soweto, Gauteng
  - Local Institution, Cape Town, Western Cape
  - Local Institution, Stellenbosch, Western Cape
- South Korea (3):
  - Local Institution, Daejeon
  - Local Institution, Incheon
  - Local Institution, Seoul
- Spain (3):
  - Hosp Univer 12 De Octubre, Madrid
  - Hospital Carlos Haya De Malaga, Málaga
  - Hospital Meixoeiro, Vigo
- Taiwan (4):
  - Local Institution, Kaohsiung City
  - Local Institution, Taichung
  - Local Institution, Taipei
  - Local Institution, Taoyuan District

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 730 participants were enrolled and 349 were randomized. 3 were randomized but not treated.Of the 381 who were not randomized,3 had an adverse event, 16 withdrew consent, 1 was lost to follow-up, 339 did not meet study entry criteria and 22 due to other reasons.
Groups:
- Experimental: 12.5mg SC BMS-931699 Weekly: Subjects received 12.5 mg SC injection of lulizumab pegol weekly.
- Experimental: 12.5mg SC BMS-931699 Every Other Week: Subjects received 12.5 mg SC injection of lulizumab pegol EOW.
- Experimental: 5mg SC Injection BMS-931699 Every Other Week: Subjects received 5 mg SC injection of lulizumab pegol EOW.
- Experimental: 1.25mg SCBMS-931699 Every Other Week: Subjects received 1.25 mg lulizumab pegol SC injection EOW
- Placebo Comparator: 0mg SC Weekly BMS-931699: Subjects received 0 milligram (mg) subcutaneous (SC) injection of matching placebo weekly.
Period: Overall Study
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Started | 69 | 68 | 68 | 70 | 71
Completed | 49 | 53 | 51 | 47 | 58
Not Completed | 20 | 15 | 17 | 23 | 13
Not completed — Poor/Non-compliance | 1 | 1 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 2 | 0
Not completed — Participant request to discontinue | 2 | 2 | 2 | 0 | 0
Not completed — Adverse Event | 8 | 4 | 9 | 8 | 2
Not completed — Lack of Efficacy | 2 | 4 | 3 | 4 | 5
Not completed — Reason not provided by Investigator | 1 | 0 | 0 | 2 | 0
Not completed — Administrative reason by sponsor | 3 | 2 | 2 | 3 | 3
Not completed — Subject no longer meets study criteria | 0 | 0 | 0 | 0 | 1
Not completed — Pregnancy | 1 | 2 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699 | Total
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71 | 346
Age, Continuous [Mean (Full Range); unit: Years] — Population: All randomized and treated participants
  Years | 41.0 [18 to 64] | 39.1 [19 to 68] | 41.9 [19 to 69] | 38.0 [19 to 69] | 40.6 [18 to 68] | 40.2 [18 to 69]
Sex/Gender, Customized [Number; unit: Participants] — Population: All randomized and treated participants
  Participants
    Females <= 50 years: number analyzed (Participants) | 67 | 66 | 65 | 66 | 65 | 329
    Females <= 50 years | 47 | 57 | 47 | 55 | 51 | 257
    Females > 50 years: number analyzed (Participants) | 67 | 66 | 65 | 66 | 65 | 329
    Females > 50 years | 20 | 9 | 18 | 11 | 14 | 72
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 66 | 65 | 66 | 65 | 329
  Male | 2 | 2 | 3 | 4 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 3 | 6 | 3 | 17
  Not Hispanic or Latino | 6 | 9 | 9 | 7 | 5 | 36
  Unknown or Not Reported | 60 | 57 | 56 | 57 | 63 | 293
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 0 | 2
  Asian | 9 | 7 | 10 | 9 | 8 | 43
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 9 | 7 | 7 | 12 | 41
  White | 38 | 46 | 41 | 43 | 41 | 209
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 16 | 6 | 9 | 10 | 10 | 51

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve a BICLA Response (BICLA Response Rate) at Day 169
Description: The British Isles Lupus Assessment Group (BILAG)-based Composite Lupus Assessment (BICLA) is a measure of systemic lupus erythematosus (SLE) response. BICLA is defined as: British Isle Lupus Assessment Group improvement, defined as BILAG As at Baseline improved to B/C/D, and BILAG Bs at baseline improved to C/D, and no BILAG worsening in other BILAG organ systems such that there are no new BILAG As or greater than 1 new BILAG B; and no worsening in the SLEDAI-2K total score compared to Baseline (defined as no increase in SLEDAI total score); and no worsening in the physician's global assessment (MDGA) of disease activity ("no worsening" is defined as less than 10% worsening, equivalent to a 10mm increase on a 100mm visual analog scale [VAS]) compared to Baseline.
Time Frame: At Day 169
Population: All Randomized and Treated participants
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Percentage of participants | 59.4 [49.7 to 69.1] | 63.2 [53.6 to 72.9] | 57.4 [47.5 to 67.2] | 58.6 [48.9 to 68.3] | 59.2 [49.6 to 68.8]
Statistical Analysis 1: Comparison: Experimental: 12.5mg SC BMS-931699 Weekly vs Placebo Comparator: 0mg SC Weekly BMS-931699; Test type: Superiority; p = 0.9745, Chi-squared; Nominal p-values that are not adjusted for multiplicity
Statistical Analysis 2: Comparison: Experimental: 12.5mg SC BMS-931699 Every Other Week vs Placebo Comparator: 0mg SC Weekly BMS-931699; Test type: Superiority; p = 0.6217, Chi-squared; Nominal p-values that are not adjusted for multiplicity
Statistical Analysis 3: Comparison: Experimental: 5mg SC Injection BMS-931699 Every Other Week vs Placebo Comparator: 0mg SC Weekly BMS-931699; Test type: Superiority; p = 0.8295, Chi-squared; Nominal p-values that are not adjusted for multiplicity
Statistical Analysis 4: Comparison: Experimental: 1.25mg SCBMS-931699 Every Other Week vs Placebo Comparator: 0mg SC Weekly BMS-931699; Test type: Superiority; p = 0.9439, Chi-squared; Nominal p-values that are not adjusted for multiplicity

2. Secondary Outcome: Percentage of Participants Who Meet Response Criteria for the SLE Responder Index : SRI(4), SRI(5) and SRI(6) at Day 169
Description: SRI is the Systemic Lupus Erythematosus Responder Index. An SRI(4) Response is defined as a reduction in Day 1 SLEDAI-2K disease activity score of ≥ 4 points AND (a)no worsening in the physician's global assessment (MDGA) of disease activity ("no worsening" is defined as less than 10% worsening, equivalent to a 10mm increase on a 100mm visual analog scale [VAS]) compared to Baseline) AND (b) no new BILAG-2004 Index A organ system score AND (c)no more than one new or worsening BILAG-2004 Index B organ system scores.
  An SRI(5) Response is defined as a reduction in Day 1 SLEDAI-2K disease activity score of ≥ 5 points AND (a) AND (b) AND (c).
  An SRI(6) Response is defined as a reduction in Day 1 SLEDAI-2K disease activity score of ≥ 6 points AND (a) AND (b) AND (c) The outcomes are better in increasing order from SRI(4) to SRI(5) to SRI(6)
Time Frame: At Day 169
Population: All randomized and treated participants
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Percentage of participants
  SRI (4) | 55.1 [45.2 to 64.9] | 48.5 [38.6 to 58.5] | 39.7 [29.9 to 49.5] | 44.3 [34.5 to 54.1] | 49.3 [39.5 to 59.1]
  SRI (5) | 37.7 [28.1 to 47.3] | 29.4 [20.3 to 38.5] | 27.9 [19.0 to 36.9] | 31.4 [22.3 to 40.6] | 33.8 [24.6 to 43.0]
  SRI (6) | 37.7 [28.1 to 47.3] | 26.5 [17.7 to 35.3] | 27.9 [19.0 to 36.9] | 31.4 [22.3 to 40.6] | 33.8 [24.6 to 43.0]

3. Secondary Outcome: Percentage of Participants Who Meet Response Criteria for the SLE Responder Index: SRI(4), SRI(5) and SRI(6) at Day 85
Description: as for outcome 2
Time Frame: At Day 85
Population: All Randomized and Treated participants
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Percentage of participants
  SRI (4) | 49.3 [39.4 to 59.2] | 48.5 [38.6 to 58.5] | 41.2 [31.4 to 51.0] | 47.1 [37.3 to 57.0] | 43.7 [34.0 to 53.3]
  SRI (5) | 29.0 [20.0 to 38.0] | 32.4 [23.0 to 41.7] | 25.0 [16.4 to 33.6] | 31.4 [22.3 to 40.6] | 28.2 [19.4 to 36.9]
  SRI (6) | 29.0 [20.0 to 38.0] | 30.9 [21.7 to 40.1] | 25.0 [16.4 to 33.6] | 31.4 [22.3 to 40.6] | 26.8 [18.1 to 35.4]

4. Secondary Outcome: Percentage of Participants With BICLA Response (BICLA Response Rate) at Day 85
Description: BICLA is defined as: British Isle Lupus Assessment Group improvement, defined as BILAG As at Baseline improved to B/C/D, and BILAG Bs at baseline improved to C/D, and no BILAG worsening in other BILAG organ systems such that there are no new BILAG As or greater than 1 new BILAG B; and no worsening in the SLEDAI-2K total score compared to Baseline (defined as no increase in SLEDAI total score); and no worsening in the physician's global assessment (MDGA) of disease activity ("no worsening" is defined as less than 10% worsening, equivalent to a 10mm increase on a 100mm visual analog scale [VAS]) compared to Baseline; No changes in concomitant medications according to the following criteria: No increase of or addition of a new immunosuppressant agent (azathioprine,mycophenolic acid/mycophenolate mofetil, methotrexate, anti-malarial, leflunomide) over baseline levels; No increase in corticosteroid dose above baseline level outside of those allowed per protocol.
Time Frame: At Day 85
Population: All Randomized and Treated Participants
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Percentage of participants | 69.6 [60.5 to 78.7] | 64.7 [55.2 to 74.2] | 57.4 [47.5 to 67.2] | 57.1 [47.4 to 66.9] | 54.9 [45.2 to 64.6]

5. Secondary Outcome: Mean Change From Baseline in CLASI Score at Day 85 and Day 169
Description: Mean change from baseline, CLASI = Cutaneous Lupus Erythematosus Disease Area and Severity Index. Scores can range from 0 to 70 with higher scores denoting greater disease activity or damage.
Time Frame: At Day 85 and Day 169
Population: All Randomized and Treated Subjects
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Scores on a scale
  Day 85: number analyzed (Participants) | 61 | 64 | 58 | 61 | 66
  Day 85 | -2.31 (3.107) | -3.20 (4.718) | -1.69 (2.319) | -1.82 (4.515) | -3.11 (4.239)
  Day 169: number analyzed (Participants) | 52 | 54 | 51 | 51 | 61
  Day 169 | -3.17 (4.387) | -3.78 (5.555) | -2.47 (2.824) | -2.94 (4.897) | -3.57 (4.177)

6. Secondary Outcome: Percentage of Participants With an Improvement of >4 or a Decrease of >50% From Baseline in Their Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) Score
Description: as for outcome 5
Time Frame: At Day 85 and Day 169
Population: All randomized and treated participants
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Percentage of participants | 39.3 [29.1 to 49.6] | 46.9 [36.6 to 57.1] | 34.5 [24.2 to 44.7] | 36.1 [26.0 to 46.2] | 42.4 [32.4 to 52.4]

7. Secondary Outcome: Change From Baseline in Arthritis, as Assessed by American College of Rheumatology (ACR) 28-joint Count of Tender and Swollen Joints on Day 85 and Day 169
Description: Mean Change from Baseline Over Time; Measured by Disease Activity Score 28: A single score on a continuous scale (0-9.4). The level of RA disease activity can be interpreted as low (DAS28 <=3.2),moderate (3.2 < DAS28 <=5.1), or as high disease activity (DAS28 > 5.1)
Time Frame: At baseline, Day 85 and Day 169
Population: All Randomized and Treated Participants
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Scores on a scale | -4.63 (4.719) | -4.63 (5.311) | -4.75 (4.985) | -4.42 (5.626) | -3.84 (4.922)

8. Secondary Outcome: Change From Baseline in BILAG-2004 Score of Systemic Lupus Erythematosus (SLE) Activity on Day 85 and Day 169
Description: Overall British Isles Lupus Assessment Group-2004 score, BILAG Scores: A=Severe disease activity, B=Moderate disease activity, C=Mild disease, D=Inactive disease but previously affected, E=System never involved.The categories are converted to a numeric score (A=9, B=3, C=1, D=0, E=0) and treated as a continuous variable. Higher score= more severe disease activity.
Time Frame: At baseline, Day 85 and Day 169
Population: All randomized and treated participants
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Score
  BILAG-2004 Score Day 85: number analyzed (Participants) | 62 | 64 | 57 | 59 | 64
  BILAG-2004 Score Day 85 | -10.31 (7.480) | -8.83 (7.749) | -7.07 (7.299) | -8.66 (6.598) | -7.94 (8.008)
  BILAG-2004 Score Day 169: number analyzed (Participants) | 52 | 54 | 51 | 51 | 58
  BILAG-2004 Score Day 169 | -11.50 (6.983) | -10.46 (7.808) | -8.98 (6.719) | -9.73 (5.478) | -9.78 (7.590)

9. Secondary Outcome: Cumulative Corticosteroid and Immunosuppressant Use
Description: Percent of participants requiring use of corticosteroids and mmunosuppressants use over time
Time Frame: Up to one day prior to the first dose of long-term extension period or up to 42 days post last short-term dose date, which ever is earlier
Population: All randomized and treated participants
Measure: Number; unit: Percentage of participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Percentage of participants
  Corticosteroids: Oral | 89.9 | 82.4 | 86.8 | 84.3 | 94.4
  Corticosteroids: Oral inhalation | 0 | 0 | 1.5 | 0 | 0
  Immunosuppressant | 46.4 | 63.2 | 38.2 | 51.4 | 59.2
  Immunosuppressant Azathioprine | 23.2 | 29.4 | 14.7 | 28.6 | 33.8
  Immunosuppressant Methotrexate | 26.1 | 35.3 | 25.0 | 24.3 | 26.8

10. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and Pre-established Events of Special Interest
Description: Although there are no identified risks for BMS-931699, BMS has developed a list of events of special interest for the BMS-931699 program based on the known biologic class effects, the mechanism of action of BMS-931699, overall potential consequences of mmunosuppression, and preliminary data from unblinded clinical trials. Event categories of special interest for this study may include, but are not limited to: Infections, Autoimmunity, Malignancies, Injection-related reactions
Time Frame: On or after the first dose date of short-term study medication and up to 42 days post last short-term dose date or up to the day prior to the first dose of long-term extension period, whichever is earlier
Population: All treated subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Participants
  Serious Adverse Events | 5 | 5 | 9 | 8 | 6
  Related SAEs | 3 | 3 | 5 | 0 | 1
  Related Adverse Events | 33 | 30 | 29 | 19 | 19
  AEs of Malignancies | 0 | 0 | 0 | 0 | 0
  AEs of Infections and Infestations | 38 | 41 | 35 | 39 | 30
  AEs Leading to Discontinuation | 8 | 5 | 9 | 9 | 3
  Adverse Events of Autoimmunity | 4 | 0 | 0 | 0 | 1
  Most Common Adverse Events | 59 | 56 | 60 | 59 | 62
  Adverse Events of Local Injection Reactions | 10 | 8 | 10 | 3 | 4

11. Secondary Outcome: Percentage of Participants With Clinically Significant Changes in Vital Signs:Heart Rate
Description: HEART RATE (HR) Beats per min (BPM): HR > 100 AND CHANGE FROM BASELINE > 30 OR HR < 55 AND CHANGE FROM BASELINE < -15
Time Frame: At Day 85 and Day 169
Population: All Treated participants
Measure: Number; unit: Percentage of participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Percentage of participants
  HEART RATE (BPM) SITTING | 5.9 | 2.9 | 2.9 | 2.9 | 5.6
  HEART RATE (BPM) STANDING | 5.9 | 4.3 | 7.4 | 7.1 | 5.7
  HEART RATE (BPM) SUPINE | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Percentage of Participants With Clinically Significant Changes in Vital Signs: Systolic and Diastolic Blood Pressure
Description: SYSTOLIC BLOOD PRESSURE (SYSBP) (MMHG); SYSBP > 140 AND CHANGE FROM BASELINE > 20 OR SYSBP < 90 AND CHANGE FROM BASELINE < -20; DIASTOLIC BLOOD PRESSURE (DIABP) > 90 AND CHANGE FROM BASELINE > 10 OR DIABP < 55 AND CHANGE FROM BASELINE < -10;
Time Frame: At Day 85 and Day 169
Population: All Treated participants
Measure: Number; unit: Percentage of participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Percentage of participants
  SYSTOLIC BLOOD PRESSURE (MMHG) SITTING | 17.6 | 11.6 | 10.3 | 10.0 | 15.5
  SYSTOLIC BLOOD PRESSURE (MMHG) STANDING | 14.7 | 14.5 | 8.8 | 11.4 | 20.0
  SYSTOLIC BLOOD PRESSURE (MMHG) SUPINE | 0 | 0 | 1 | 0 | 0
  DIASTOLIC BLOOD PRESSURE (MM HG) SITTING | 17.6 | 26.1 | 11.8 | 17.1 | 9.9
  DIASTOLIC BLOOD PRESSURE (MM HG) STANDING | 27.9 | 18.8 | 25.0 | 21.4 | 20.0
  DIASTOLIC BLOOD PRESSURE (MM HG) SUPINE | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Percentage of Participants With Clinically Significant Changes in Vital Signs: Respiration Rate
Description: RESPIRATION RATE (RESP) (PER MIN) RESP > 16 OR RESP CHANGE FROM BASELINE > 10
Time Frame: At Day 85 and Day 169
Population: All Treated participants
Measure: Number; unit: Percentage of participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Percentage of participants | 82.4 | 85.5 | 75.0 | 70.0 | 81.7

14. Secondary Outcome: Percentage of Participants With Clinically Significant Changes in Vital Signs: Temperature
Description: TEMPERATURE (TEMP) (C) TEMP > 38.3 OR TEMP CHANGE FROM BASELINE > 1.6
Time Frame: At Day 85 and Day 169
Population: All Treated participants
Measure: Number; unit: Percentage of participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Percentage of participants | 0 | 0 | 1.5 | 1.4 | 1.4

15. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: QTc (corrected QT) Fridericia, PR Interval, QRS Interval and Change from baseline in QTCF
Time Frame: Up to 42 days post last dose of short-term double-blind study medication or up to the day prior to the start of long-term extension period, whichever is earlier.
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Participants
  QTC Fredericia (msec) <= 450 | 56 | 58 | 58 | 56 | 65
  QTC Fredericia (msec) 450< To <= 480 | 12 | 8 | 5 | 11 | 5
  QTC Fredericia (msec) 480 < to <= 500 | 0 | 1 | 2 | 0 | 1
  QTC Fredericia (msec) > 500 | 1 | 1 | 3 | 3 | 0
  PR Interval (msec) <= 200 | 69 | 68 | 64 | 66 | 68
  PR Interval (msec) > 200 | 0 | 0 | 4 | 4 | 3
  QRS Interval (msec) <= 120 | 68 | 67 | 66 | 67 | 70
  QRS Interval (msec) > 120 | 1 | 1 | 2 | 3 | 1
  Change from baseline in QTCF (msec) <= 30: number analyzed (Participants) | 68 | 68 | 64 | 60 | 67
  Change from baseline in QTCF (msec) <= 30 | 66 | 59 | 54 | 55 | 62
  Change from baseline in QTCF (msec) 30 To <= 60: number analyzed (Participants) | 68 | 68 | 64 | 60 | 67
  Change from baseline in QTCF (msec) 30 To <= 60 | 2 | 7 | 7 | 2 | 5
  Change from baseline in QTCF (msec) > 60: number analyzed (Participants) | 68 | 68 | 64 | 60 | 67
  Change from baseline in QTCF (msec) > 60 | 0 | 2 | 3 | 3 | 0

16. Secondary Outcome: Ctrough: Trough Level Serum Concentration of BMS-931699 at Time Point Specified
Description: Pharmacokinetics of BMS-931699 derived from serum concentration versus time data; Ctrough = Trough level serum concentration of BMS-931699 at time point specified Pharmacokinetic Population: defined as all subjects who receive any study medication and have any available concentration-time data.
Time Frame: Day 169
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 68 | 68 | 68 | 70 | 71
ng/mL | 2040 (945.57) | 640.8 (436.35) | 207.1 (149.53) | 62.2 (56.83) | 0 (0)

17. Secondary Outcome: Serum Biomarkers C3, C4
Description: Serum biomarkers C3, C4, anti-double-stranded deoxyribonucleic acid (anti-dsDNA), anti-nuclear antibody (ANA) and other autoantibodies were measured from blood serum samples collected on Day 85 and Day 169
Time Frame: At Day 85 and Day 169
Population: All Treated participants with at Least One Post-Treatment Biomarker Measurement
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
g/L
  C3, Baseline: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  C3, Baseline | 1.068 (0.3405) | 1.029 (0.3265) | 0.990 (0.3318) | 1.028 (0.3149) | 0.991 (0.2641)
  C3, Day 85: number analyzed (Participants) | 62 | 64 | 58 | 61 | 66
  C3, Day 85 | 1.037 (0.3024) | 1.014 (0.3428) | 1.030 (0.3225) | 1.083 (0.3124) | 0.986 (0.3005)
  C3, Day 169: number analyzed (Participants) | 53 | 54 | 55 | 51 | 58
  C3, Day 169 | 1.045 (0.3405) | 1.010 (0.3557) | 1.027 (0.3528) | 1.077 (0.3256) | 0.992 (0.2981)
  C4, Baseline: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  C4, Baseline | 0.201 (0.1084) | 0.185 (0.1088) | 0.177 (0.0861) | 0.202 (0.0984) | 0.183 (0.0824)
  C4, Day 85: number analyzed (Participants) | 62 | 64 | 58 | 61 | 66
  C4, Day 85 | 0.206 (0.1037) | 0.195 (0.1079) | 0.190 (0.0875) | 0.215 (0.0965) | 0.179 (0.0824)
  C4, Day 169: number analyzed (Participants) | 53 | 54 | 55 | 51 | 58
  C4, Day 169 | 0.212 (0.1161) | 0.185 (0.1014) | 0.187 (0.0941) | 0.207 (0.0927) | 0.184 (0.0896)

18. Secondary Outcome: Serum Biomarkers: Anti-Nuclear Antibodies (ANA)
Description: Serum biomarkers C3, C4, anti-double-stranded deoxyribonucleic acid (anti-dsDNA), anti-nuclear antibody (ANA) and other autoantibodies were measured from blood serum samples collected on Day 85 and Day 169. No anti-dsDNA data was available for this report
Time Frame: At Day 85 and Day 169
Population: All Treated participants with at Least One Post-Treatment Biomarker Measurement
Measure: Number; unit: Percentage
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 66 | 67 | 70
Percentage
  Baseline Negative Day 85 Negative: number analyzed (Participants) | 9 | 7 | 2 | 8 | 5
  Baseline Negative Day 85 Negative | 62.5 | 57.1 | 100.0 | 50.0 | 60.0
  Baseline Negative Day 85 Positive: number analyzed (Participants) | 9 | 7 | 2 | 8 | 5
  Baseline Negative Day 85 Positive | 37.5 | 42.9 | 0 | 50.0 | 40.0
  Baseline Positive Day 85 Negative: number analyzed (Participants) | 53 | 58 | 55 | 51 | 62
  Baseline Positive Day 85 Negative | 11.3 | 3.4 | 1.8 | 2.0 | 0
  Baseline Positive Day 85 Positive: number analyzed (Participants) | 53 | 58 | 55 | 51 | 62
  Baseline Positive Day 85 Positive | 88.7 | 96.6 | 98.2 | 98.0 | 100.0
  Baseline Negative Day 169 Negative: number analyzed (Participants) | 7 | 6 | 3 | 7 | 5
  Baseline Negative Day 169 Negative | 71.4 | 33.3 | 100.0 | 57.1 | 40.0
  Baseline Negative Day 169 Positive: number analyzed (Participants) | 7 | 6 | 3 | 7 | 5
  Baseline Negative Day 169 Positive | 28.6 | 66.7 | 0 | 42.9 | 60.0
  Baseline Positive Day 169 Negative: number analyzed (Participants) | 43 | 51 | 52 | 47 | 56
  Baseline Positive Day 169 Negative | 9.3 | 2.0 | 5.8 | 4.3 | 1.8
  Baseline Positive Day 169 Positive: number analyzed (Participants) | 43 | 51 | 52 | 47 | 56
  Baseline Positive Day 169 Positive | 90.7 | 98.0 | 94.2 | 95.7 | 98.2

19. Secondary Outcome: Short Term: Receptor Occupancy Over Time
Description: Percent CD4+ Receptor Occupancy and percent CD8+ Receptor Occupancy
Time Frame: At Day 85 and Day 169
Population: All Treated participants with at Least One Post-Treatment Biomarker Measurement
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 66 | 67 | 71
Percentage
  %CD4+ RO Baseline: number analyzed (Participants) | 54 | 54 | 54 | 51 | 54
  %CD4+ RO Baseline | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  %CD4+ RO Day 85: number analyzed (Participants) | 44 | 48 | 45 | 42 | 41
  %CD4+ RO Day 85 | 95.722 (12.1298) | 83.244 (28.9616) | 70.520 (32.9107) | 37.155 (31.2927) | 0.350 (0.5997)
  %CD4+ RO Day 169: number analyzed (Participants) | 32 | 39 | 37 | 33 | 36
  %CD4+ RO Day 169 | 92.390 (22.1377) | 77.210 (29.3976) | 74.286 (28.5105) | 44.115 (34.3707) | 0.334 (0.4460)
  %CD8+ RO Baseline: number analyzed (Participants) | 57 | 58 | 56 | 57 | 57
  %CD8+ RO Baseline | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  %CD8+ RO Day 85: number analyzed (Participants) | 47 | 52 | 47 | 47 | 45
  %CD8+ RO Day 85 | 95.831 (7.6571) | 81.730 (30.4345) | 68.960 (32.0543) | 32.516 (29.7242) | 0.160 (0.3120)
  %CD8+ RO Day 169: number analyzed (Participants) | 35 | 41 | 37 | 35 | 39
  %CD8+ RO Day 169 | 92.043 (20.6963) | 74.726 (33.0060) | 69.850 (30.5880) | 40.989 (31.9867) | 0.235 (0.5438)

20. Secondary Outcome: Percentage of Participants With BMS-931699 Induced Antibody Response Over Time Point Specified
Description: Immunogenicity defined as positive for anti-drug antibodies post-baseline measurement if baseline missing or negative. If baseline is positive, then immunogenicity is defined as a positive post-baseline measurement with titer value 4 times greater than baseline. (A) all subjects with a laboratory reported positive antibody responses to BMS-931699 during the short-term double-blind treatment period are included. Overall: At least one positive sample relative to baseline during short-term double-blind and follow-up period.
Time Frame: Day 169
Population: All Treated participants with at Least One Post-Treatment Immunogenicity Assessment Who Developed Laboratory Reported Positive Antibody Responses to BMS-931699
Measure: Number; unit: Percentage of participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 41 | 34 | 34 | 26 | 0
Percentage of participants
  % with Neutralizing activity | 23.1 | 41.2 | 64.7 | 34.1 |
  % with Neutralizing activity (Baseline) | 0 | 5.9 | 0 | 0 |
  % with Neutralizing activity (Overall) | 23.1 | 35.3 | 64.7 | 34.1 |

21. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in General Laboratory Tests: HEMATOLOGY I
Description: HEMATOLOGY I: ERYTHROCYTE/PLATELET ATTRIBUTES HEMOGLOBIN G/L L < 0.85×PRE-RX; HEMATOCRIT VOL L < 0.85×PRE-RX; PLATELET COUNT X10*9 C/L H > 1.5×ULN (ULN = Upper Limit of Normal) IF PRE-RX IS MISSING OR > 1.5×ULN PLATELET COUNT X10*9 C/L L < 0.85×LLN (LLN = Lower Limit of Normal) IF PRE-RX IS MISSING OR < 0.85×LLN IF PRE-RX >= LLN OR < 0.85×PRE-RX IF PRE-RX < LLN; ERYTHROCYTES RBC X10*12 C/L L < 0.85×PRE-RX HEMATOLOGY II QUANTITATIVE WBC : LEUKOCYTES X10*9 C/L H > 1.2×ULN IF PRE-RX IS MISSING OR > 1.2×ULN IF LLN <= PRE-RX <= ULN OR > 1.5×PRE-RX IF PRE-RX > ULN OR > ULN IF PRE-RX < LLN; LEUKOCYTES WBC X10*9 C/L L < 0.9×LLN IF PRE-RX IS MISSING OR < 0.9×LLN IF LLN <= PRE-RX <= ULN OR < 0.85×PRE-RX IF PRE-RX < LLN OR < LLN IF PRE-RX > ULN
Time Frame: Up to 42 days post last dose of study medication in short-term or long-term extension period
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Participants
  Erythrocytes Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Erythrocytes Low | 4 | 4 | 6 | 3 | 5
  Erythrocytes High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Erythrocytes High | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Hematocrit Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Hematocrit Low | 6 | 10 | 5 | 5 | 8
  Hematocrit High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Hematocrit High | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Hemoglobin Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Hemoglobin Low | 4 | 4 | 5 | 4 | 5
  Hemoglobin High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Hemoglobin High | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Platelet count low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Platelet count low | 1 | 1 | 1 | 1 | 2
  Platelet count high: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Platelet count high | 0 | 0 | 0 | 1 | 0
  Quantitative WBC: Leukocytes low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Quantitative WBC: Leukocytes low | 12 | 18 | 12 | 16 | 16
  Quantitative WBC: Leukocytes high: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Quantitative WBC: Leukocytes high | 1 | 1 | 0 | 3 | 1

22. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in General Laboratory Tests: HEMATOLOGY II
Description: WBC DIFFERENTIAL COUNT: BASOPHILS (ABSOLUTE) X10*9 C/L H > 0.4; BLASTS (ABSOLUTE) X10*9 C/L H > 0; EOSINOPHILS (ABSOLUTE) EOSA X10*9 C/L H > 0.75; LYMPHOCYTES (ABSOLUTE) X10*9 C/L H > 7.5; LYMPHOCYTES (ABSOLUTE) X10*9 C/L L < 0.75; MONOCYTES (ABSOLUTE) X10*9 C/L H > 2; NEUTROPHILS (ABSOLUTE) X10*9 C/L L < 1.5 IF PRE-RX IS MISSING OR < 1.5 IF PRE-RX >= 1.5 OR < 0.85×PRE-RX IF PRE-RX < 1.5; COAGULATION activated Partial thromboplastin time (APTT) SEC H > 1.5×ULN; INTL NORMALIZED RATIO (INR) INR FRACTION H > 1.5×ULN PROTHROMBIN TIME (PT) PT SEC H > 1.5×ULN
Time Frame: Up to 42 days post last dose of study medication in short-term or long-term extension period
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Participants
  Basophils (Absolute) Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Basophils (Absolute) Low | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Basophils (Absolute) High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Basophils (Absolute) High | 0 | 0 | 0 | 0 | 0
  Blasts (Absolute) Low: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Blasts (Absolute) Low |  | NA — Not evaluated |  |  |
  Blasts (Absolute) High: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Blasts (Absolute) High |  | 0 |  |  |
  Eosinophils (Absolute) Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Eosinophils (Absolute) Low | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Eosinophils (Absolute) High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Eosinophils (Absolute) High | 3 | 0 | 0 | 2 | 1
  Lymphocytes (Absolute) Low | 21 | 29 | 24 | 25 | 25
  Lymphocytes (Absolute) High | 0 | 0 | 0 | 0 | 0
  Monocytes (Absolute) High | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Monocytes (Absolute) Low | 0 | 0 | 0 | 0 | 0
  Neutrophils (Absolute) Low | 10 | 8 | 5 | 7 | 4
  Neutrophils (Absolute) High | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated

23. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in General Laboratory Tests : LIVER FUNCTION TESTS
Description: LIVER FUNCTION TESTS:ALKALINE PHOSPHATASE (ALP) ALP U/L H > 1.25×ULN IF PRE-RX IS MISSING OR > 1.25×ULN IF PRE-RX <= ULN OR > 1.25×PRE-RX IF PRE-RX > ULN; ALANINE AMINOTRANSFERASE (ALT) ALT U/L H > 1.25×ULN IF PRE-RX IS MISSING OR > 1.25×ULN IF PRE-RX <= ULN OR > 1.25×PRE-RX IF PRE-RX > ULN; ASPARTATE AMINOTRANSFERASE (AST) AST U/L H > 1.25×ULN IF PRE-RX IS MISSING OR > 1.25×ULN IF PRE-RX <= ULN OR > 1.25×PRE-RX IF PRE-RX > ULN; BILIRUBIN, DIRECT UMOL/L H > 1.1×ULN IF PRE-RX IS MISSING OR > 1.1×ULN IF PRE-RX <= ULN OR > 1.25×PRE-RX IF PRE-RX > ULN G-GLUTAMYL TRANSFERASE (GGT) GGT U/L H > 1.15×ULN IF PRE-RX IS MISSING OR > 1.15×ULN IF PRE-RX <= ULN OR > 1.2×PRE-RX IF PRE-RX > ULN BILIRUBIN, TOTAL UMOL/L H > 1.1×ULN IF PRE-RX IS MISSING OR > 1.1×ULN IF PRE-RX <= ULN OR > 1.25×PRE-RX IF PRE-RX > ULN
Time Frame: Up to 42 days post last dose of study medication in short-term or long-term extension period
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Participants
  Alanine Aminotransferase Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Alanine Aminotransferase Low | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Alanine Aminotransferase High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Alanine Aminotransferase High | 12 | 17 | 6 | 9 | 8
  Alkaline Phosphatase Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Alkaline Phosphatase Low | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Alkaline Phosphatase High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Alkaline Phosphatase High | 2 | 3 | 2 | 5 | 8
  Aspartate Aminotransferase Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Aspartate Aminotransferase Low | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Aspartate Aminotransferase High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Aspartate Aminotransferase High | 10 | 13 | 11 | 8 | 10
  Bilirubin, Direct Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Bilirubin, Direct Low | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Bilirubin Direct, High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Bilirubin Direct, High | 0 | 13 | 0 | 1 | 0
  Bilirubin Total, Low | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Bilirubin Total, High | 0 | 0 | 0 | 1 | 1
  G-Glutamyl Transferase, Low: number analyzed (Participants) | 69 | 68 | 68 | 68 | 71
  G-Glutamyl Transferase, Low | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  G-Glutamyl Transferase, High: number analyzed (Participants) | 69 | 68 | 68 | 68 | 71
  G-Glutamyl Transferase, High | 18 | 14 | 16 | 15 | 13

24. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in General Laboratory Tests: KIDNEY FUNCTION TESTS
Description: KIDNEY FUNCTION TESTS:BLOOD UREA NITROGEN MMOL/L H > 1.1×ULN IF PRE-RX IS MISSING OR > 1.1×ULN IF PRE-RX <= ULN OR > 1.2×PRE-RX IF PRE-RX > ULN CREATININE UMOL/L H > 1.5×ULN IF PRE-RX IS MISSING OR > 1.5×ULN IF PRE-RX <= ULN OR > 1.33×PRE-RX IF PRE-RX > ULN GLOMERULAR FILTRATION RATE, CALC. ML/S/M*2 L < 0.8×PRE-RX; UREA UREA MMOL/L H > 1.1×ULN IF PRE-RX IS MISSING OR > 1.1×ULN IF PRE-RX <= ULN OR > 1.2×PRE-RX IF PRE-RX > ULN
Time Frame: Up to 42 days post last dose of study medication in short-term or long-term extension period
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Participants
  Blood Urea Nitrogen, Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Blood Urea Nitrogen, Low | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Blood Urea Nitrogen, High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Blood Urea Nitrogen, High | 9 | 11 | 3 | 14 | 10
  Creatinine, Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Creatinine, Low | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Creatinine, High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Creatinine, High | 2 | 0 | 0 | 2 | 1
  GLOMERULAR FILTRATION RATE, CALC. Low: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  GLOMERULAR FILTRATION RATE, CALC. Low |  |  | 0 |  |
  GLOMERULAR FILTRATION RATE, CALC. High: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  GLOMERULAR FILTRATION RATE, CALC. High |  |  | NA — Not evaluated |  |
  Urea, Low: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0
  Urea, Low | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated |
  Urea, High: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0
  Urea, High | 0 | 0 | 0 | 0 |

25. Secondary Outcome: Number of Participants Clinically Significant Abnormalities in General Laboratory Tests ELECTROLYTES 1
Description: CALCIUM, TOTAL MMOL/L H > 1.1×ULN IF PRE-RX IS MISSING OR > 1.1×ULN IF PRE-RX <= ULN OR > 1.1×PRE-RX IF PRE-RX > ULN OR > ULN IF PRE-RX < LLN; CALCIUM, TOTAL MMOL/L L < 0.9×LLN IF PRE-RX IS MISSING OR < 0.9×LLN IF PRE-RX >= LLN OR < 0.9×PRE-RX IF PRE-RX < LLN OR < LLN IF PRE-RX > ULN; CHLORIDE, SERUM MMOL/L H > 1.1×ULN IF PRE-RX IS MISSING OR > 1.1×ULN IF PRE-RX <= ULN OR > 1.1×PRE-RX IF PRE-RX > ULN OR > ULN IF PRE-RX < LLN; CHLORIDE, SERUM MMOL/L L < 0.9×LLN IF PRE-RX IS MISSING OR < 0.9×LLN IF PRE-RX >= LLN OR < 0.9×PRE-RX IF PRE-RX < LLN OR < LLN IF PRE-RX > ULN;
Time Frame: Up to 42 days post last dose of study medication in short-term or long-term extension period
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Participants
  Calcium, Total, Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Calcium, Total, Low | 0 | 0 | 1 | 0 | 0
  Calcium, Total, High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Calcium, Total, High | 0 | 0 | 0 | 0 | 0
  Chloride, Serum, Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Chloride, Serum, Low | 0 | 0 | 0 | 0 | 0
  Chloride, Serum, High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Chloride, Serum, High | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Number of Participants Clinically Significant Abnormalities in General Laboratory Tests: ELECTROLYTES 2
Description: BICARBONATE MMOL/L H > 1.2×ULN IF PRE-RX IS MISSING OR > 1.2×ULN IF PRE-RX <= ULN OR > 1.2×PRE-RX IF PRE-RX > ULN OR > ULN IF PRE-RX < LLN; BICARBONATE MMOL/L L < 0.8×LLN IF PRE-RX IS MISSING OR < 0.8×LLN IF PRE-RX >= LLN OR < 0.8×PRE-RX IF PRE-RX < LLN OR < LLN IF PRE-RX > ULN; POTASSIUM, SERUM MMOL/L H > 1.1×ULN IF PRE-RX IS MISSING OR > 1.1×ULN IF PRE-RX <= ULN OR > 1.1×PRE-RX IF PRE-RX > ULN OR > ULN IF PRE-RX < LLN; POTASSIUM, SERUM MMOL/L L < 0.9×LLN IF PRE-RX IS MISSING OR < 0.9×LLN IF PRE-RX >= LLN OR < 0.9×PRE-RX IF PRE-RX < LLN OR < LLN IF PRE-RX > ULN; MAGNESIUM, SERUM MMOL/L H > 1.1×ULN IF PRE-RX IS MISSING OR > 1.1×ULN IF PRE-RX <= ULN OR > 1.1×PRE-RX IF PRE-RX > ULN OR > ULN IF PRE-RX < LLN MAGNESIUM, SERUM MMOL/L L < 0.9×LLN IF PRE-RX IS MISSING OR < 0.9×LLN IF PRE-RX >= LLN OR < 0.9×PRE-RX IF PRE-RX < LLN OR < LLN IF PRE-RX > ULN
Time Frame: Up to 42 days post last dose of study medication in short-term or long-term extension period
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Participants
  Bicarbonate, Low: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0
  Bicarbonate, Low |  |  | 0 |  |
  Bicarbonate, High: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0
  Bicarbonate, High |  |  | 0 |  |
  Magnesium, Serum, Low: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Magnesium, Serum, Low |  |  | 0 |  |
  Magnesium, Serum, High: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Magnesium, Serum, High |  |  | 0 |  |
  Potassium, Serum, Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Potassium, Serum, Low | 1 | 0 | 1 | 1 | 1
  Potassium, Serum, High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Potassium, Serum, High | 0 | 0 | 1 | 1 | 0

27. Secondary Outcome: Number of Participants Clinically Significant Abnormalities in General Laboratory Tests: ELECTROLYTES 3
Description: SODIUM, SERUM MMOL/L H > 1.05×ULN IF PRE-RX IS MISSING OR > 1.05×ULN IF PRE-RX <= ULN OR > 1.05×PRE-RX IF PRE-RX > ULN OR > ULN IF PRE-RX < LLN SODIUM, SERUM MMOL/L L < 0.95×LLN IF PRE-RX IS MISSING OR < 0.95×LLN IF PRE-RX >= LLN OR < 0.95×PRE-RX IF PRE-RX < LLN OR < LLN IF PRE-RX > ULN PHOSPHORUS, INORGANIC PHOS MMOL/L H > 1.25×ULN IF PRE-RX IS MISSING OR > 1.25×ULN IF PRE-RX <= ULN OR > 1.25×PRE-RX IF PRE-RX > ULN OR > ULN IF PRE-RX < LLN PHOSPHORUS, INORGANIC PHOS MMOL/L L < 0.85×LLN IF PRE-RX IS MISSING OR < 0.85×LLN IF PRE-RX >=LLN OR < 0.85×PRE-RX IF PRE-RX < LLN OR < LLN IF PRE-RX > ULN
Time Frame: Up to 42 days post last dose of study medication in short-term or long-term extension period
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Participants
  Sodium, Serum Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Sodium, Serum Low | 0 | 0 | 0 | 0 | 0
  Sodium, Serum High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Sodium, Serum High | 0 | 0 | 0 | 0 | 0
  Phosphorus, Inorganic, Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Phosphorus, Inorganic, Low | 0 | 2 | 4 | 1 | 0
  Phosphorus, Inorganic, High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Phosphorus, Inorganic, High | 0 | 0 | 0 | 1 | 0

28. Secondary Outcome: Number of Participants Clinically Significant Abnormalities in General Laboratory Tests : OTHER CHEMISTRY TESTING 1
Description: GLUCOSE TESTS:GLUCOSE, FASTING SERUM MMOL/L H > 1.3×ULN IF PRE-RX IS MISSING OR > 1.3×ULN IF PRE-RX <= ULN OR > 2×PRE-RX IF PRE-RX > ULN OR > ULN IF PRE-RX < LLN GLUCOSE, FASTING SERUM MMOL/L L < 0.8×LLN IF PRE-RX IS MISSING OR < 0.8×LLN IF PRE-RX >= LLN OR < 0.8×PRE-RX IF PRE-RX < LLN OR < LLN IF PRE-RX > ULN; PROTEIN TESTS:ALBUMIN G/L L < 0.9×LLN IF PRE-RX IS MISSING OR < 0.9×LLN IF PRE-RX >= LLN OR < 0.9×PRE-RX IF PRE-RX < LLN PROTEIN, TOTAL G/L H > 1.1×ULN IF PRE-RX IS MISSING OR > 1.1×ULN IF PRE-RX <= ULN OR > 1.1×PRE-RX IF PRE-RX > ULN OR > ULN IF PRE-RX < LLN PROTEIN, TOTAL G/L L < 0.9×LLN IF PRE-RX IS MISSING OR < 0.9×LLN IF PRE-RX >= LLN OR < 0.9×PRE-RX IF PRE-RX < LLN OR < LLN IF PRE-RX > ULN
Time Frame: Up to 42 days post last dose of study medication in short-term or long-term extension period
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Participants
  Glucose, Fasting serum, Low: number analyzed (Participants) | 69 | 67 | 65 | 68 | 71
  Glucose, Fasting serum, Low | 1 | 3 | 0 | 4 | 5
  Glucose, Fasting Serum, High: number analyzed (Participants) | 69 | 67 | 67 | 68 | 71
  Glucose, Fasting Serum, High | 3 | 3 | 0 | 0 | 4
  Albumin, Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Albumin, Low | 1 | 2 | 2 | 2 | 1
  Albumin, High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 41
  Albumin, High | 0 | 0 | 0 | 0 | 0
  Protein, Total, Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Protein, Total, Low | 0 | 0 | 1 | 1 | 0
  Protein, Total, High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Protein, Total, High | 0 | 0 | 1 | 1 | 0

29. Secondary Outcome: Number of Participants Clinically Significant Abnormalities in General Laboratory Tests : OTHER CHEMISTRY TESTING 2
Description: OTHER CHEMISTRY TESTING LIPID TESTS: CHOLESTEROL, TOTAL (TC) MMOL/L H > 1.2×ULN IF PRE-RX IS MISSING OR > 1.2×ULN IF PRE-RX <= ULN OR > 1.2×PRE-RX IF PRE-RX > ULN TRIGLYCERIDES, FASTING MMOL/L H > 1.25×ULN IF PRE-RX IS MISSING OR > 1.25×ULN IF PRE-RX <= ULN OR > 1.5×PRE-RX IF PRE-RX > ULN PANCREATIC TESTS: AMYLASE, TOTAL U/L H > 1.5×ULN; LIPASE, TOTAL (TURBIDIMETRIC ASSAY) U/L H > 1.5×ULN; LIPASE, TOTAL (COLORIMETRIC ASSAY) U/L H > 1.5×ULN; ENDOCRINE TESTS:CORTISOL, AM NMOL/L L < 138 THYROID STIMULATING HORMONE (TSH) TSH MU/L H > 1.5×ULN IF PRE-RX IS MISSING OR > 1.5×ULN IF PRE-RX <= ULN OR > 2×PRE-RX IF PRE-RX > ULN
Time Frame: Up to 42 days post last dose of study medication in short-term or long-term extension period
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Participants
  Cholesterol, Total (TC) Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Cholesterol, Total (TC) Low | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Cholesterol, Total (TC) High: number analyzed (Participants) | 69 | 68 | 65 | 68 | 71
  Cholesterol, Total (TC) High | 5 | 4 | 12 | 10 | 8
  Triglycerides, Fasting Low: number analyzed (Participants) | 69 | 67 | 67 | 68 | 71
  Triglycerides, Fasting Low | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Triglycerides, Fasting High: number analyzed (Participants) | 69 | 67 | 65 | 68 | 71
  Triglycerides, Fasting High | 12 | 13 | 12 | 10 | 8
  Amylase, Total Low: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0
  Amylase, Total Low |  |  | NA — Not evaluated |  |
  Amylase, Total High: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0
  Amylase, Total High |  |  | 0 |  |
  Lipase, Total (Colorimetric Assay) Low: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0
  Lipase, Total (Colorimetric Assay) Low |  |  | NA — Not evaluated |  |
  Lipase, Total (Colorimetric Assay) High: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0
  Lipase, Total (Colorimetric Assay) High |  |  | 1 |  |
  Lipase, Total (Turbidimetric Assay) Low: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Lipase, Total (Turbidimetric Assay) Low |  |  | NA — Not evaluated |  |
  Lipase, Total (Turbidimetric Assay) High: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Lipase, Total (Turbidimetric Assay) High |  |  | 1 |  |
  Thyroid Stimulating Hormone, Low: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Thyroid Stimulating Hormone, Low |  |  | NA — Not evaluated |  |
  Thyroid Stimulating Hormone, High: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Thyroid Stimulating Hormone, High |  |  | 0 |  |

30. Secondary Outcome: Number of Participants Clinically Significant Abnormalities in General Laboratory Tests : OTHER CHEMISTRY TESTING 3
Description: OTHER CHEMISTRY TESTING CARDIAC TESTS: CREATINE KINASE (CK) CK U/L H > 1.5×ULN IF PRE-RX IS MISSING OR > 1.5×ULN IF PRE-RX <= ULN OR > 1.5×PRE-RX IF PRE-RX > ULN; TROPONIN-I, CARDIAC SPECIFIC UG/L H > ULN; METABOLITE TESTS:URIC ACID URIC MMOL/L H > 1.2×ULN IF PRE-RX IS MISSING OR > 1.2×ULN IF PRE-RX <= ULN OR > 1.25×PRE-RX IF PRE-RX > ULN; CHEM TEST, MULTI INDICATIONS : LACTATE DEHYDROGENASE (LD) LD U/L H > 1.25×ULN IF PRE-RX IS MISSING OR > 1.25×ULN IF PRE-RX <= ULN OR > 1.5×PRE-RX IF PRE-RX > ULN
Time Frame: Up to 42 days post last dose of study medication in short-term or long-term extension period
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Participants
  Creatine Kinase Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Creatine Kinase Low | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Creatine Kinase High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Creatine Kinase High | 5 | 5 | 3 | 3 | 1
  TROPONIN-I, CARDIAC SPECIFIC Low: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  TROPONIN-I, CARDIAC SPECIFIC Low |  |  | NA — Not evaluated |  |
  TROPONIN-I, CARDIAC SPECIFIC High: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  TROPONIN-I, CARDIAC SPECIFIC High |  |  | 0 |  |
  Uric Acid, Low: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0
  Uric Acid, Low |  |  | NA — Not evaluated |  |
  Uric Acid, High: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0
  Uric Acid, High |  |  | 0 |  |
  Lactate dehydrogenase (LD) low: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Lactate dehydrogenase (LD) low |  |  | NA — Not evaluated |  |
  Lactate dehydrogenase (LD) high: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Lactate dehydrogenase (LD) high |  |  | 0 |  |

31. Secondary Outcome: Number of Participants Clinically Significant Abnormalities in General Laboratory Tests : IMMUNOLOGY
Description: IMMUNE ACTIVATION MARKERS:C-REACTIVE PROTEIN (CRP) CRP MG/L H > 1.5×ULN; CRP, HIGH SENSITIVITY MG/L H > 1.5×ULN;
Time Frame: Up to 42 days post last dose of study medication in short-term or long-term extension period
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Participants
  C-Reactive Protein (CRP) Low: number analyzed (Participants) | 68 | 68 | 65 | 64 | 69
  C-Reactive Protein (CRP) Low | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  C-Reactive Protein (CRP) High: number analyzed (Participants) | 68 | 68 | 65 | 64 | 69
  C-Reactive Protein (CRP) High | 19 | 18 | 22 | 18 | 22
  CRP, High Sensitivity Low: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
  CRP, High Sensitivity Low |  |  | NA — Not evaluated | NA — Not evaluated |
  CRP, High Senstivity High: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
  CRP, High Senstivity High |  |  | 1 | 0 |

32. Secondary Outcome: Number of Participants Clinically Significant Abnormalities in General Laboratory Tests : URINALYSIS
Description: QUALITATIVE URINE CHEMISTRY: BLOOD, URINE N/A H >= 2 IF PRE-RX IS MISSING OR >= 2 IF PRE-RX < 1 OR >= 2×PRE-RX IF PRE-RX >= 1 GLUCOSE, URINE N/A H >= 1 IF PRE-RX IS MISSING OR >= 1 IF PRE-RX < 1 OR >= 2×PRE-RX IF PRE-RX >= 1 PROTEIN, URINE UNKNOWN H >= 2 IF PRE-RX IS MISSING OR >= 2 IF PRE-RX < 1 OR >= 2×PRE-RX IF PRE-RX >= 1 URINALYSIS II URINE WBC + RBC ; RBC, URINE HPF H >= 2 IF PRE-RX IS MISSING OR >= 2 IF PRE-RX < 2 OR >= 4 IF PRE-RX >= 2 WBC, URINE HPF H >= 2 IF PRE-RX IS MISSING OR >= 2 IF PRE-RX < 2 OR >= 4 IF PRE-RX >= 2
Time Frame: Up to 42 days post last dose of study medication in short-term or long-term extension period
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Participants
  Blood, Urine, Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Blood, Urine, Low | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Blood, Urine, High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Blood, Urine, High | 18 | 21 | 20 | 21 | 20
  Glucose, Urine, Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Glucose, Urine, Low | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Glucose, Urine, High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Glucose, Urine, High | 2 | 2 | 0 | 0 | 1
  Protein, Urine, Low: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Protein, Urine, Low | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  Protein, Urine, High: number analyzed (Participants) | 69 | 68 | 67 | 68 | 71
  Protein, Urine, High | 7 | 7 | 13 | 7 | 10
  RBC, Urine, Low: number analyzed (Participants) | 54 | 56 | 54 | 47 | 50
  RBC, Urine, Low | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  RBC, Urine, High: number analyzed (Participants) | 54 | 56 | 54 | 47 | 50
  RBC, Urine, High | 18 | 19 | 13 | 17 | 18
  WBC, Urine, Low: number analyzed (Participants) | 65 | 64 | 62 | 65 | 65
  WBC, Urine, Low | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated | NA — Not evaluated
  WBC, Urine, High: number analyzed (Participants) | 65 | 64 | 62 | 65 | 65
  WBC, Urine, High | 28 | 29 | 31 | 31 | 25

33. Secondary Outcome: Change From Baseline in the SLEDAI-2K Score of SLE Activity on Day 85 and Day 169
Description: Systemic Lupus Erythematosus Disease Activity Index, SLEDAI; Version 2000, also known as SLEDAI-2K. The SLEDAI-2K score is a weighted, cumulative index of lupus disease activity. SLEDAI-2K is calculated from 24 individual descriptors across 9 organ systems; 0 indicates inactive disease and the maximum theoretical score is 105.
Time Frame: At baseline, Day 85 and Day 169
Population: All randomized and treated participants
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Score
  SLEDAI-2K Score Day 85: number analyzed (Participants) | 62 | 63 | 58 | 61 | 66
  SLEDAI-2K Score Day 85 | -3.61 (3.345) | -3.24 (3.320) | -3.17 (3.304) | -4.02 (3.960) | -3.29 (3.953)
  SLEDAI-2K Score Day 169: number analyzed (Participants) | 52 | 54 | 51 | 51 | 61
  SLEDAI-2K Score Day 169 | -4.88 (3.370) | -4.17 (4.064) | -3.98 (3.478) | -4.82 (4.078) | -4.15 (3.728)

34. Secondary Outcome: Change From Baseline in Physician Global Assessment of Disease Activity (MDGA) on Day 85 and Day 169
Description: Physician Global Assessment of Arthritis was measured by asking the physician to assess the participant's current arthritis disease activity by placing a vertical line on a 0 to 100 millimeter (mm) visual analog scale (VAS), where 0 mm = very good and 100 mm = very bad.
Time Frame: At baseline, Day 85 and Day 169
Population: All randomized and treated participants
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Experimental: 12.5mg SC BMS-931699 Weekly | Experimental: 12.5mg SC BMS-931699 Every Other Week | Experimental: 5mg SC Injection BMS-931699 Every Other Week | Experimental: 1.25mg SCBMS-931699 Every Other Week | Placebo Comparator: 0mg SC Weekly BMS-931699
Number analyzed (Participants) | 69 | 68 | 68 | 70 | 71
Score
  MDGA score Day 85: number analyzed (Participants) | 62 | 64 | 58 | 60 | 65
  MDGA score Day 85 | -28.77 (18.193) | -23.87 (20.321) | -21.00 (20.596) | -20.55 (17.233) | -23.83 (20.752)
  MDGA score Day 169: number analyzed (Participants) | 69 | 53 | 68 | 50 | 71
  MDGA score Day 169 | -29.30 (17.371) | -26.87 (21.284) | -28.68 (19.919) | -26.71 (18.182) | -25.28 (19.952)

ADVERSE EVENTS:
Time Frame: All non-serious adverse events (NSAEs) and serious adverse events (SAEs) are reported from onset on or after the first dose date of study medication and up to 42 days post last dose.
Groups:
- Placebo - Short Term (ST): Subjects received 0 milligram (mg) subcutaneous (SC) injection of matching placebo weekly.
- Lulizumab Pegol 12.5 mg Weekly - ST: Subjects received 12.5 mg SC injection of lulizumab pegol weekly.
- Lulizumab Pegol 12.5 mg EOW - ST: Subjects received 12.5 mg SC injection of lulizumab pegol EOW.
- Lulizumab Pegol 5 mg EOW - ST: Subjects received 5 mg SC injection of lulizumab pegol EOW.
- Lulizumab Pegol 1.25 mg Every Other Week (EOW) - ST: Subjects received 1.25 mg lulizumab pegol SC injection EOW.
Arm/Group | Placebo - Short Term (ST) | Lulizumab Pegol 12.5 mg Weekly - ST | Lulizumab Pegol 12.5 mg EOW - ST | Lulizumab Pegol 5 mg EOW - ST | Lulizumab Pegol 1.25 mg Every Other Week (EOW) - ST
All-Cause Mortality (participants affected / at risk) | 0/71 | 2/69 | 0/68 | 0/68 | 0/70
Serious Adverse Events (participants affected / at risk) | 6/71 | 5/69 | 5/68 | 9/68 | 8/70
Other Adverse Events (participants affected / at risk) | 41/71 | 45/69 | 43/68 | 47/68 | 39/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Short Term (ST) (N=71) | Lulizumab Pegol 12.5 mg Weekly - ST (N=69) | Lulizumab Pegol 12.5 mg EOW - ST (N=68) | Lulizumab Pegol 5 mg EOW - ST (N=68) | Lulizumab Pegol 1.25 mg Every Other Week (EOW) - ST (N=70)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Lupus enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Serum sickness (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 3 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Zika virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 2
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Putamen haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Lupus nephritis (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Short Term (ST) (N=71) | Lulizumab Pegol 12.5 mg Weekly - ST (N=69) | Lulizumab Pegol 12.5 mg EOW - ST (N=68) | Lulizumab Pegol 5 mg EOW - ST (N=68) | Lulizumab Pegol 1.25 mg Every Other Week (EOW) - ST (N=70)
Leukopenia (Blood and lymphatic system disorders) | 0 | 5 | 3 | 3 | 3
Lymphopenia (Blood and lymphatic system disorders) | 0 | 4 | 4 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 11 | 7 | 1 | 5 | 5
Nausea (Gastrointestinal disorders) | 4 | 5 | 0 | 5 | 5
Chest pain (General disorders) | 4 | 1 | 1 | 2 | 1
Injection site pain (General disorders) | 4 | 2 | 3 | 4 | 2
Injection site reaction (General disorders) | 0 | 4 | 2 | 3 | 0
Pyrexia (General disorders) | 2 | 1 | 1 | 3 | 4
Bronchitis (Infections and infestations) | 3 | 4 | 1 | 3 | 1
Gastroenteritis (Infections and infestations) | 1 | 8 | 3 | 2 | 1
Influenza (Infections and infestations) | 2 | 0 | 4 | 3 | 2
Nasopharyngitis (Infections and infestations) | 5 | 9 | 4 | 8 | 6
Pharyngitis (Infections and infestations) | 4 | 2 | 5 | 7 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 7 | 3 | 8 | 8
Urinary tract infection (Infections and infestations) | 3 | 6 | 11 | 9 | 11
Vaginal infection (Infections and infestations) | 1 | 2 | 5 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 4 | 3 | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 4 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 1 | 4
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2 | 3 | 1
Dizziness (Nervous system disorders) | 3 | 3 | 3 | 1 | 5
Headache (Nervous system disorders) | 9 | 10 | 9 | 7 | 5
Migraine (Nervous system disorders) | 2 | 0 | 1 | 4 | 1
Depression (Psychiatric disorders) | 0 | 0 | 4 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 2 | 3 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2015-05-03): https://cdn.clinicaltrials.gov/large-docs/44/NCT02265744/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-28): https://cdn.clinicaltrials.gov/large-docs/44/NCT02265744/SAP_001.pdf